CLINICAL TRIAL: NCT06196606
Title: Effect of Botulinum Toxin Injection Into Upper Esophageal Sphincter on Swallowing Function in Patients With Medullary Infarction
Brief Title: Effect of Botulinum Toxin Injection Into Upper Esophageal Sphincter in Patients With Medullary Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yuli Zhu, postgraduate, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-0297-002
Record Dates: First submitted 2023-12-22; First posted 2024-01-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Brain Stem Infarctions; Dysphagia, Oropharyngeal; Dysphagia, Esophageal
Keywords: Botulinum Toxins; Esophageal Sphincter, Upper
MeSH Terms: conditions — Brain Stem Infarctions; Deglutition Disorders | interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Botulinum toxin type A for injection (Hengli National Drug approval number S10970037) 100U, diluted with 1 ml.9% sodium chloride solution for reserve use.Each patient was injected with 90U
  Interventions: Drug: Botulinum toxin type A for injection

INTERVENTIONS:
Drug: Botulinum toxin type A for injection — Botulinum toxin was injected into the upper esophageal sphincter of each patient
  Other Names: Botulinum toxin type A for injection (Hengli National Drug approval number S10970037)

SUMMARY:
Dysphagia is an important complication in patients with medullary infarction, the incidence rate is 57%-69%. Compared with other brain infarctions, the medulla oblongata involves multiple swallowing-related nerve nuclei, and the possibility of brain remodeling after injury is small. Dysphagia has become a prominent clinical problem in patients with medullary infarction, which can lead to malnutrition, decrease the quality of life of patients and affect the prognosis of the disease. Solving this clinical problem is particularly important for patients with medullary infarction. The incidence of UES opening disorder in patients with medullary infarction is as high as 80%, and the clinical problem of UES opening disorder is enthusiastically studied at home and abroad. At present, the intervention measures include balloon dilatation, surgical incision and botulinum toxin injection. Balloon dilatation is easy to cause mucosal edema and damage, and cricopharyngeal myotomy often has complications such as local infection, massive hemorrhage and local nerve injury. There is no significant difference between the success rate of UES botulinum toxin injection and surgical incision. Among the above measures, UES botulinum toxin injection has a good clinical application prospect, but the drug dosage and injection method are still not unified in clinic. In particular, how to accurately locate has become a hot topic in current research. On this basis, this study uses ultrasound combined with balloon localization to inject UES botulinum toxin and make clinical observation.

DETAILED DESCRIPTION:
Under the ultrasound combined with balloon fixation, two injection sites were selected from the left upper esophageal sphincter, and 30U was injected respectively, and one injection site was selected from the right side, and 30U was injected. In addition, the patient also received routine swallowing training once a day for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* MRI examination of the head confirmed the medullary infarction.
* Those who have not significantly improved swallowing function after standardized rehabilitation treatment for more than 2 weeks (FOIS remains unchanged or decreases)
* Video-fluroscopic swallowing study (VFSS) indicated incomplete/non-opening of the cricopharyngeal muscle
* Based on Fiberoptic endoscopic evaluation of swallowing, the hyoid bone moves upward more than half the height of the C3 cone
* Vital signs are stable
* The patient himself or his family voluntarily signed a written informed consent form.

Exclusion Criteria:

* Brain MRI showed that there were lesions in other areas outside the medulla oblongata
* People who have suffered from stroke in the past
* Patients with severe cognitive impairment, mental illness and severe cardiopulmonary disease
* Abnormal throat structure
* Malignant tumor patient
* Patients with other neuromuscular diseases
* Infection or wound at the injection site
* Botulinum toxin allergic person
* Hemorrhagic tendency and coagulation dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Functional Oral Intake Scale | day 1 ，day 14，day28 and day 180
  According to whether the patient can eat by mouth and the degree of dependence on nasal feeding tube, it is divided into 7 grades, corresponding to 1-7 points respectively. The higher the score, the better the swallowing function.
Rosenbek penetration-aspiration scale | day 1 and day 14
  Based on the results of Videofluroscopic swallowing study (VFSS), the cases of leakage and aspiration were divided into 8 grades, corresponding to 1-8 points respectively. The higher the score, the better the swallowing function.

SECONDARY OUTCOMES:
Murray secretion scale | day 1 and day 14
  Based on Fiberoptic endoscopic evaluation of swallowing (FEES), the accumulation position of oropharyngeal secretions was described and divided into 4 grades. The higher the score, the worse the swallowing function.
yale pharyngeal residue severity rating scale | day 1 and day 14
  Based on Fiberoptic endoscopic evaluation of swallowing (FEES), the main indicators include the location of the residue (epiglottic valley and pyriform sinus) and the amount of residue, which is divided into 5 grades. The higher the score, the worse the swallowing function.
fiberoptic endoscopic dysphagia severity scale | day 1 and day 14
  Based on Fiberoptic endoscopic evaluation of swallowing (FEES), Eat different foods and observe whether penetration aspiration and protective reflex occur. The highest score is 6, which means that saliva accumulates with penetration or aspiration, and the lowest score is 1. When eating soft solid food, there is no leakage or aspiration, and there is little or moderate residue in epiglottic valley or pyriform sinus. The higher the score, the worse the swallowing function.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No
Due to the privacy policy of the First Affiliated Hospital of Zhengzhou University, the data cannot be disclosed, but it can be obtained from the PI with an appropriate reason